CLINICAL TRIAL: NCT03698617
Title: A Phase IIa, Open-label, Propofol-controlled ,Dose-escalation, Multi-center Study to Evaluate the Tolerance, Efficacy and Safety of HSK3486 for Induction of General Anesthesia in Elective Surgery Patients.
Brief Title: A Phase IIa Study Investigating the Tolerance, Efficacy and Safety of HSK3486
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-202
Record Dates: First submitted 2018-09-18; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Induction of General Anaesthesia
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): Dose Escalation Cohort:
  0.1 mg/kg, 0.2 mg/kg, 0.3mg/kg 0.4 mg/kg 0.5 mg/kg, 0.6 mg/kg, 0.7mg/kg, 0.8 mg/kg Dose Expansion Cohort: 0.3 mg/kg and 0.5 mg/kg.
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): Dose Escalation Cohorts:2.0mg/kg and 2.5mg/kg; Dose Expansion Cohorts: 2.0mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — For induction of general anesthesia In dose escalation cohort: Starting from 0.4mg/kg, up-titration dose by 0.1mg/kg until 0.8mg//kg or down-titration dose by 0.1mg/kg until 0.1mg/kg based on the efficacy and safety results.
  Arms: HSK3486
Drug: Propofol — For induction of general anesthesia
  Arms: Propofol

SUMMARY:
This is a Phase IIa, open-label, propofol-controlled ,dose-escalation, multi-center Study to evaluate the tolerance, efficacy and safety of HSK3486 for induction of general anesthesia in elective surgery patients.This study is consisted of two cohorts, dose-escalation and dose-expansion cohorts. The doses in dose- expansion cohort were selected from dose-escalation results.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients required tracheal intubation under general anesthesia and a non-emergency non-cardiothoracic and non-extracranial elective surgery for an estimated duration of ≤ 3 h ;.
2. Males or females, aged ≥ 18 and ≤ 65 years old;
3. Body mass index (BMI) ≥ 19 and ≤ 30 kg/m2;
4. ASA grade I~II;
5. Capable of understanding the procedure and method of this study, willing to sign an informed consent form and to complete this study in strict accordance with the study protocol.

Exclusion Criteria:

1. Patients were contraindicated in general anesthesia.;
2. Patients with a known sensitivity to propofol, opioids, naloxone, eggs, soy products or a medical condition such that these agents were contraindicated
3. Patients in receipt of any investigational drug within 30 days before screening.
4. Patients in receipt of propofol, opioid , other sedative or anesthetic or analgesics within one month prior to the screening period.
5. Patients in receipt of general anesthesia surgery within two weeks prior to the screening period.
6. The patient has some history or evidence of increased risk of sedation or anesthesia, such as cardiovascular disease, respiratory disease, cerebrovascular disease, liver, kidney, blood system, or metabolic system disease prior to the screening period.
7. Abnormal laboratory results consisting of any of the following: :

1) AST and ALT≥ 2×ULN； 2）TBIL≥ 1.5×ULN； 3）Hb≤ 90g/L; 4）ANC≤1.5×109/L; 5) PLT≤80×109/L； 6） serum creatinine≥ 1.5×ULN.

8. Patients with a history of drug or ethanol abuse with the past 3 months. 9. Pregnant women or female patients with a positive serum or urine human chorionic gonadotropin pregnancy test at screening or baseline or lactating female patients. . 10. 10. Patients with a positive Allen 's test who collected arterial blood for PK study.

11. Patients with respiratory management difficulties. 12. Patients with an inability to communicate well with the investigator, or deemed unsuitable according to the investigator (in each case providing a reason).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
The success rate of induction of general anesthesia | during induction of general anesthesia on day 1
  To find the MTD or the RP2D of HSK3486 in the induction of general anesthesia, the success rate of induction of general anesthesia is the primary outcome measurement.

SECONDARY OUTCOMES:
Time from start of IMP administration to loss of eyelash reflex | during induction of general anesthesia on day 1
Time from start of IMP administration to loss of consciousness | during induction of general anesthesia on day 1
Time from start of IMP administration to intubation and the intubation reaction | during induction of general anesthesia on day 1
Mini-Mental State Examination (MMSE) total scores(0-30) by time point | Pre-dose to 48 hours post-dose
  Change from baseline in Mini-Mental State Examination (MMSE) total score
change from baseline in blood pressure （systolic, diastolic and mean arterial pressure) | pre-dose to 20 minutes post-dose
  safety endpoits
change from baseline in heart rate | pre-dose to 20 minutes post-dose
  safety endpoits
change from baseline in arterial oxygen saturation | pre-dose to 20 minutes post-dose
  safety endpoits
Number of patients with adverse events | Pre-dose to 48 hours post-dose
  safety endpoits

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Affiliated Hospital of WMU, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhu Q, Luo Z, Wang X, Wang D, Li J, Wei X, Tang J, Yao S, Ouyang W, Zhang W, Zuo Y, Wang X, Liu J. Efficacy and safety of ciprofol versus propofol for the induction of anesthesia in adult patients: a multicenter phase 2a clinical trial. Int J Clin Pharm. 2023 Apr;45(2):473-482. doi: 10.1007/s11096-022-01529-x. Epub 2023 Jan 21. PMID 36680620